CLINICAL TRIAL: NCT06633016
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of ABX-002 for the Adjunctive Treatment of Major Depressive Disorder
Brief Title: Study of ABX-002 for the Adjunctive Treatment of Major Depressive Disorder (AMPLIFY)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Autobahn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABX-002-2001
Record Dates: First submitted 2024-09-30; First posted 2024-10-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study participants, Investigator, and study site staff, Sponsor will be blinded to treatment assignments (ABX-002 or placebo solution).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABX-002 + SSRI/SNRI (Experimental): Patients continue to receive their selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study in addition to ABX-002.
  Interventions: Drug: ABX-002
- Placebo + SSRI/SNRI (Placebo Comparator): Patients continue to receive their selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study in addition to the Placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ABX-002 — ABX-002 oral solution in 1-mL cyclic olefin polymer prefilled syringes, taken on an empty stomach first thing in the morning followed by 240 mL (8 oz) of water.
  Arms: ABX-002 + SSRI/SNRI
Other: Placebo — Comparator Placebo oral solution in 1-mL cyclic olefin polymer prefilled syringes, taken on an empty stomach first thing in the morning followed by 240 mL (8 oz) of water.
  Arms: Placebo + SSRI/SNRI

SUMMARY:
The goal of this clinical trial is to learn if ABX-002 added to an existing antidepressant treatment will benefit depression symptoms in adults with moderate to severe major depressive disorder who have had an inadequate response to their antidepressant.

This is a double-blind, placebo-controlled, 2-arm, parallel-group, Phase 2 study, randomized 1:1 (ABX-002: placebo).

The study will include the following stages:

1. Screening, approximately 35 days
2. 42-day Treatment Period
3. 2-week post dose Safety Follow-up Period
4. 6-month postdose targeted safety follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Meets the DSM-5 criteria for Major Depressive Disorder, with a current major depressive episode duration of > 6 weeks and ≤ 18 months.
* A score of ≤ 22 (midrange mild/moderate) on the Hamilton Anxiety Rating Scale.
* Montgomery-Asberg Depression Rating Scale total score of > 24 [indicating moderate to severe depression] at Screening and at Baseline.
* Subject is compliantly using a single selective serotonin reuptake inhibitors / serotonin norepinephrine reuptake inhibitor antidepressant for at least 6 weeks for their current episode of depression, with an adequate dose, and with an inadequate response as defined by the Antidepressant Treatment Response Questionnaire. The dosage of the current antidepressant must have been stable for the past 4 weeks, and the dosage and specific antidepressant used should remain the same from Screening through the end of the Follow-up Period.

Exclusion Criteria:

Note: History implies lifetime history, unless otherwise specified

* History of schizophrenia or other psychotic disorder, major depressive disorder with psychotic features or concomitant DSM-5 depressive disorders, bipolar I or II disorder, cyclothymic disorder, delirium, dementia, amnestic disorder, or cognitive disorder.
* Current diagnosis or active symptoms within the last 2 years of obsessive-compulsive disorder, posttraumatic stress disorder, panic disorder, or eating disorder, according to DSM-5 criteria.
* Primary diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder, according to DSM-5 criteria. Current or history within the last 2 years of self-injurious behavior is exclusionary.
* Has failed more than 2 single selective serotonin reuptake inhibitors / serotonin norepinephrine reuptake inhibitor antidepressant treatments, including the current serotonin reuptake inhibitors / serotonin norepinephrine reuptake inhibitor, during the current depressive episode, despite an adequate dose (per Antidepressant Treatment Response Questionnaire) and duration (at least 6 weeks).
* Failure to respond to triiodothyronine or thyroxine augmentation for the treatment of depression.
* Started new psychotherapy or had a change in the intensity of psychotherapy within 8 weeks before Screening.
* Is suicidal at Screening or Baseline
* History or current evidence within previous 3 months before Screening of uncontrolled, clinically significant neurological, gastrointestinal, respiratory, renal, hepatic, immunological, hematological, or other medical disorder, including cancer, that would jeopardize the safe participation of the subject in the study (in the opinion of the Investigator).
* History of thyroid disease
* History of multiple endocrine neoplasia syndrome
* Diagnosis of epilepsy or history of convulsions, including childhood febrile seizure. Use of co-administered drugs that may lower seizure threshold is excluded.
* Females who are pregnant, intend to become pregnant or are breastfeeding.
* Antidepressants: Prior use of psychedelics, ketamine, or esketamine, for the treatment of Major Depressive Disorder.
* Antidepressants: Current use, or use within 4 weeks prior to Screening, of any other augmentation agents for Major Depressive Disorder (e.g. second-generation antipsychotics [SGA], monoamine oxidase inhibitors [MAOI], tricyclic antidepressants [TCA], lithium, or bupropion)
* Current or prior use of treatment for hypothyroidism including but not limited to synthetic or natural thyroid hormone, triiodothyronine and/or thyroxine.
* Concomitant use of biotin of any dose and in any preparation 14 days prior to Day 1 until after the last study visit at Week 8 (Day 56).
* Medications that are strong cytochrome P450 3A4 inhibitors or strong cytochrome P450 3A4 inducers are not allowed.
* Prescription drug/controlled substance abuse, or illicit substance use within 1 year of Screening or positive urine drug results at Screening or Baseline for an illicit substance.
* History or presence of cataract on ophthalmic examination (including slit-lamp), glaucoma, inflammatory eye disease or prior ophthalmic surgical procedures or laser surgery in either eye

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the 17-item Hamilton Rating Scale for Depression (HAMD-17) | 6 weeks
  The HAMD-17 is a clinician-based assessment of depressive symptoms. Higher scores indicate worse symptoms. A score of 0-9 is generally accepted to be within the normal range (or in clinical remission), while a score of greater than 17 indicates moderate to severe depression symptoms.

SECONDARY OUTCOMES:
Change from Baseline for Clinical Global Impression of Severity (CGI-S) | 6 weeks
  a 7-point rating scale used to measure illness and symptom severity in subjects with mental disorders. The greater the number the more severe.
Change from Baseline for Sheehan Disability Scale (SDS) | 6 weeks
  Self-rated, 3-item questionnaire that uses a Likert scale from 0 (not at all) to 10 (extremely) to assess impairment in the occupational, social, and family domains.
Change from baseline for 6-item Hamilton Rating Scale for Depression (HAMD-6) | 6 weeks
  Six-item scale used to assess the core symptoms of depression.
Change from baseline for 29-item Hamilton Rating Scale for Depression (HAMD-29) | 6 weeks
  Clinician-based assessment of depressive symptoms. HAMD-29 covers HAMD-6, HAMD-17 (items 1 to 17), the Melancholia Scale (MES) (items 18 to 23), and the neurovegetative symptoms (NVS) (items 24 to 28).
Patient Global Impression-Improvement (PGI-I) | 6 weeks
  Quality-of-life questionnaire to assess improvement of activities of daily living, wellbeing, and function.
Assessment of safety and tolerability of ABX-002 compared with placebo using adverse events | 6 weeks
  Incidence and severity of treatment-emergent adverse events to ABX-002 will be measured

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Autobahn Site #131, Birmingham, Alabama
  - Autobahn Site #132, Chandler, Arizona
  - Autobahn Site #116, Phoenix, Arizona
  - Autobahn Site #136, Tucson, Arizona
  - Autobahn Site #150, Anaheim, California
  - Autobahn Site #113, Encino, California
  - Autobahn Site #133, Encino, California
  - Autobahn Site #124, Glendale, California
  - Autobahn Site #140, Long Beach, California
  - Autobahn Site #121, Los Alamitos, California
  - Autobahn Site #117, Newport Beach, California
  - Autobahn Site #106, Oceanside, California
  - Autobahn Site #152, Orange, California
  - Autobahn Site #151, Rancho Cucamonga, California
  - Autobahn Site #119, San Jose, California
  - Autobahn Site #126, Walnut Creek, California
  - Autobahn Site #149, West Covina, California
  - Autobahn Site #122, Cromwell, Connecticut
  - Autobahn Site #108, Brandon, Florida
  - Autobahn Site #110, Hialeah, Florida
  - Autobahn Site #101, Jacksonville, Florida
  - Autobahn Site #139, Lake City, Florida
  - Autobahn Site #111, Miami, Florida
  - Autobahn Site #141, Miami, Florida
  - Autobahn Site #147, Miami Gardens, Florida
  - Autobahn Site #102, Orlando, Florida
  - Autobahn Site #148, Tampa, Florida
  - Autobahn Site #123, Atlanta, Georgia
  - Autobahn Site #112, Decatur, Georgia
  - Autobahn Site #142, Peachtree Corners, Georgia
  - Autobahn Site #120, Savannah, Georgia
  - Autobahn Site #154, Elgin, Illinois
  - Autobahn Site #137, Boston, Massachusetts
  - Autobahn Site #138, Watertown, Massachusetts
  - Autobahn Site #127, Saint Charles, Missouri
  - Autobahn Site #130, Las Vegas, Nevada
  - Autobahn Site #129, Berlin, New Jersey
  - Autobahn Site #105, Brooklyn, New York
  - Autobahn Site #134, Brooklyn, New York
  - Autobahn Site #125, New York, New York
  - Autobahn Site #104, Staten Island, New York
  - Autobahn Site #109, Beachwood, Ohio
  - Autobahn Site #107, Oklahoma City, Oklahoma
  - Autobahn Site #128, North Charleston, South Carolina
  - Autobahn Site #153, Beaumont, Texas
  - Autobahn Site #146, San Antonio, Texas
  - Autobahn Site #144, Sherman, Texas
  - Autobahn Site #159, Orem, Utah
  - Autobahn Site #145, Fairfax, Virginia
  - Autobahn Site #143, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No